CLINICAL TRIAL: NCT05773664
Title: A Phase I De-Escalation Study of Dexamethasone with Azeliragon for Management of Post-Resection Cerebral Edema in Patients with Glioblastoma
Brief Title: Dexamethasone and Azeliragon for Management of Post-Resection Cerebral Edema in Patients with Glioblastoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22367; NCI-2023-00007 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22367 (Other: City of Hope Medical Center); P30CA033572 (NIH); U19CA264512 (NIH)
Record Dates: First submitted 2023-01-30; First posted 2023-03-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Glioblastoma; Malignant Glioma
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — azeliragon; Specimen Handling; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (azeliragon, dexamethasone) (Experimental): Patients receive azeliragon PO and dexamethasone PO or IV throughout the study. Patients also undergo collection of cavity fluid and blood samples, CT scan, and brain MRI with or without contrast throughout the study.
  Interventions: Drug: Azeliragon; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast
- Arm II (dexamethasone) (Active Comparator): Patients receive dexamethasone PO or IV throughout the study. Patients also undergo collection of cavity fluid and blood samples, CT scan, and brain MRI with or without contrast throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Dexamethasone; Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast

INTERVENTIONS:
Drug: Azeliragon — Given PO
  Arms: Arm I (azeliragon, dexamethasone)
Procedure: Biospecimen Collection — Undergo collection of cavity fluid and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Procedure: Magnetic Resonance Imaging of the Brain with and without Contrast — Undergo MRI with or without contrast
  Other Names: Brain Magnetic Resonance Imaging with and without Contrast; Brain MRI; Brain MRI with and without Contrast; Head MRI with and without Contrast

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of dexamethasone when given with azeliragon in managing cerebral edema after surgery (post-resection) in patients with glioblastoma. Cerebral edema is a pathological increase in the water mass contained within the brain interstitial space. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Azeliragon is an oral RAGE inhibitor. Blocking the RAGE pathway at the time of surgery (peri-operatively) may decrease cerebral edema. Giving dexamethasone with azeliragon may help control post-operative cerebral edema in decreasing doses of concurrently administered dexamethasone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the lowest dose of dexamethasone that needs to be co-administered with azeliragon for treatment of post-resection cerebral edema in patients with glioblastoma.

II. Assess the safety of administering azeliragon peri-operatively to patients with glioblastoma.

SECONDARY OBJECTIVES:

I. Describe post-operative changes in levels of cytokines and chemokines in brain interstitium and peripheral blood in study participants.

II. Quantitatively assess changes in the volume of cerebral edema post-operatively in study participants.

III. Determine brain concentrations of azeliragon in resected tumor tissue from Arm 1 participants.

EXPLORATORY OBJECTIVES:

I. Describe post-operative changes in levels of RAGE ligands in brain interstitium, peripheral blood, and resection cavity fluid (when possible to obtain) in study participants.

II. Describe changes in levels of cytokines, chemokines, and immune cell populations in resection cavity fluid (when possible to obtain).

III. Describe differences in levels of cytokines, chemokines and RAGE ligands between patients in Arm 1 and Arm 2.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive azeliragon orally (PO) and dexamethasone PO or intravenously (IV) throughout the study. Patients also undergo collection of cavity fluid and blood samples, computed tomography (CT) scan, and brain magnetic resonance imaging (MRI) with or without contrast throughout the study.

ARM II: Patients receive dexamethasone PO or IV throughout the study. Patients also undergo collection of cavity fluid and blood samples, CT scan, and brain MRI with or without contrast throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative
* Age: >= 18 years
* Karnofsky performance status of >= 60%
* Histologically confirmed glioblastoma or radiographic findings consistent with a high grade glioma in patients undergoing surgery for initial diagnosis
* If midline shift is present on the pre-op brain MRI, it must be less than 10 mm
* The patient is planning to undergo a standard of care craniotomy, and the neurosurgeon anticipates being able to perform a gross total resection of tumor
* If a patient is taking more than 3 mg twice daily (bid) of dexamethasone at the time of signing the consent form, it is anticipated by the neurosurgeon that the participant will be able to decrease their dose of dexamethasone to 3 mg bid by 6 days before the surgery

  * Note: If the patient is not able to decrease their dose of dexamethasone to 3 mg BID 6 days before surgery, then the patient will not be allowed to participate in the study
* The patient is not planning to participate in another clinical trial during the study period
* The patient has recovered from any acute toxic effects (except alopecia) to =< grade 1 of prior anti-cancer therapy
* Absolute neutrophil count (ANC) >= 1,000/mm^3
* Platelets >= 100,000/mm^3
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease)
* Aspartate aminotransferase (AST) =< 1.5 x ULN
* Alanine aminotransferase (ALT) =< 1.5 x ULN
* Creatinine clearance of >= 60 mL/min by the Cockcroft-Gault formula
* International normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN
* Corrected QT (QTc) =< 480 ms

  * Note: To be performed within 28 days prior to day 1 of protocol therapy
* People of childbearing potential: negative urine or serum pregnancy test
* Agreement by people of childbearing potential to use an effective method of birth control or abstain from heterosexual activity for the course of the study through at least 3 months after the last dose of protocol therapy

  * Childbearing potential defined as not being surgically sterilized (regardless of gender) or not being free from menses for > 1 year (people with uteri only)

Exclusion Criteria:

* Less than 6 weeks since taking a nitrosourea-containing chemotherapy regimen; less than 4 weeks since completing a non-nitrosourea-containing cytotoxic chemotherapy regimen (except temozolomide: only patients with an interval of less than 23 days from the last dose administered when treated with the temozolomide regimen of daily for 5 days, repeated every 28 days are excluded); less than 2 weeks from taking the last dose of a targeted agent; less than 4 weeks from the last dose of bevacizumab
* Less than 3 months since focal brain radiation unless recurrent disease has been confirmed surgically or the area of recurrent tumor is outside of the radiation field
* The patient is taking a medication that is a strong CYP3A4 inducers/ inhibitors within 14 days prior to day -6 of protocol therapy
* The patient is unwilling to stop taking herbal medications prior to the start of study treatment
* The patient is taking a hepatic enzyme-inducing anticonvulsant within 14 days prior to day -6 of protocol therapy
* Clinically significant uncontrolled illness
* Active infection requiring antibiotics
* Human immunodeficiency virus (HIV)-positive
* Undergoing treatment for another cancer
* Issues with tolerating oral medication (e.g. inability to swallow pills, malabsorption issues, ongoing nausea or vomiting)
* Chronic or active viral infection of the central nervous system (CNS)
* Pregnant or breastfeeding
* Coagulopathy or bleeding disorder
* Inability to undergo a brain MRI
* Inability to tolerate dexamethasone
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-29 (Estimated); Study Completion 2024-11-29 (Estimated)

PRIMARY OUTCOMES:
Lack of feasibility | Up to 8 days after surgery
  Defined by exceeding the planned total dose of dexamethasone (per dose level) during post-operative days 1 to 8 by approximately 50%.
Incidence of adverse events | Up to 30 days post-last dose of protocol therapy
  Azeliragon related adverse events and dose limiting toxicity rate assessed per Common Terminology Criteria for Adverse Events version 5.0.

SECONDARY OUTCOMES:
Cytokines/chemokines | Up to 3 days after surgery
  Will assess cytokines/chemokines in brain interstitium and peripheral blood. The cytokine and chemokine levels will be measured as concentrations (pg/mL) and reported as a median with range.
Volume of cerebral edema | Up to 8 days after surgery
  Will assess volume of cerebral edema for each post-surgery brain magnetic resonance imaging (MRI) as measured qualitatively and quantitatively by manual segmentation and computer assisted techniques.
Azeliragon concentrations | Up to 8 days after surgery
  Will assess azeliragon concentrations in tumor samples compared to azeliragon concentrations in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Jana L Portnow, Principal Investigator — City of Hope Medical Center